CLINICAL TRIAL: NCT00565695
Title: Evaluation of the Aspheric ReSTOR IOL After Routine Cataract Extraction
Brief Title: Evaluation of the Aspheric ReSTOR Intraocular Lens (IOL) After Routine Cataract Extraction
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Kerry D. Solomon, Medcial University of South Carolina
Other Study IDs: SEI-07-002
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Cataract Extraction; Refractive Surgery
Keywords: Visual Outcomes; Patient Satisfaction; Cataract Extraction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: aspheric ReSTOR multifocal intraocular lens (IOL) — Multifocal intraocular lens

SUMMARY:
The purpose of this study is to evaluate the visual outcomes and patient satisfaction after bilateral implantation of the aspheric ReSTOR multifocal intraocular lens (IOL) and compare it to a historical control group of patients implanted bilaterally with the spherical ReSTOR multifocal IOL.

DETAILED DESCRIPTION:
Cataract is prevalent throughout the world and IOLs are routinely implanted after the extraction of the cataractous lens. It is the most frequently performed surgery in the United States with an estimated 2-3 million procedures performed annually. With the aging population on the rise, as well as the increasing popularity of refractive intraocular lenses, the number of intraocular surgeries continues to rise. Over the years, the surgical technique has evolved from intracapsular extraction to modern phacoemulsification. This development has helped with the evolution of IOLs as well. The IOLs have advanced extensively: different materials and designs are available, permitting implantation through smaller, sutureless incisions. Traditional IOLs are of monofocal design providing vision at one distance, typically far. Patients implanted with traditional monofocal IOLs usually require glasses for near distance tasks such as reading. The new multifocal IOLs offer the possibility of seeing well at more than one distance, without glasses or contacts.

The AcrySof ReSTOR (Alcon Laboratories) uses apodized diffractive technology - a design that responds to how wide or small the eye's pupil might be - to provi de near, intermediate, and distance vision. Clinical studies used to support the March 2005 FDA approval showed that 80% of people who received the lens did not use glasses for any activities after their cataract surgery; 84% who received the lens in both eyes had distance vision of 20/25 or better, with near vision of 20/32 or better. Wavefront analysis is a technique currently used to measure the aberrations of the entire optical system. The term aberration derives from the Latin ab-erratio, which means going offtrack or deviating. Therefore, and aberration is the difference that exists between the ideal image of that we would expect to see when the luminous rays are refracted in the perfect optical system (Snell's law) and what is actually achieved. This technology is widely used in refractive surgery with successful outcomes. With the introduction of wavefront analysis, a new tool is available to re-design and study the performance of IOLs. Regarding IOL design, it has been used to modify the IOL to partially compensate for the average spherical aberration. The goal is to improve the ocular optical quality of pseudophakic patients. Clinical results using the aspheric monofocal IOLs confirm that this modification leads to a significant improvement, particularly in contrast sensitivity, mesopic visual quality and reduction of high order aberrations mainly spherical aberration when compare to spherical IOLs. The new aspheric ReSTOR IOL is the first single piece acrylic multifocal IOL to be available in the United States and a comparison to a regular (spherical) multifocal IOL is necessary to determine if the aspheric ReSTOR lens shows the same improvement.

The purpose of this study is to evaluate the visual outcomes and patient satisfaction after bilateral implantation of the aspheric ReSTOR multifocal intraocular lens (IOL) and compare it to a historical control group of patients implanted bilaterally with the spherical ReSTOR multifocal IOL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects MUST fulfill the following conditions to qualify for enrollment into the trial
* Subject must have an age-related cataract in both eyes.
* 40 years of age or older.
* Patient must desire cataract extraction.
* Expected maximum of 2 weeks and minimum of 1-week interval between first and second eye surgeries.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Preoperative ocular pathology:

  * Amblyopia
  * Rubella cataract
  * Proliferative diabetic retinopathy
  * Shallow anterior chamber
  * Macular edema
  * Retinal detachment
  * Aniridia or iris atrophy
  * Uveitis
  * History of iritis
  * Iris neovascularization
  * Medically uncontrolled glaucoma
  * Microphthalmus or macrophthalmus
  * Optic nerve atrophy
  * Macular degeneration (with anticipated best postoperative visual acuity less than 20/30)
  * Advanced glaucomatous damage, etc.
* Keratometric astigmatism exceeding 1.50 diopters.
* Planned postoperative refraction for mono-vision.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device
* implantation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.
* Other ocular surgery at the time of the cataract extraction.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aspheric ReSTOR multifocal intraocular lens (IOL)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-10; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, MD, Principal Investigator — Medical University of South Carolina, Storm Eye Institute
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States